CLINICAL TRIAL: NCT05329415
Title: Tuberculosis Drug Levels and Continuous Glucose Monitoring in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: v1 20.07.2021
Record Dates: First submitted 2021-09-17; First posted 2022-04-15 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis; Diabetes Mellitus
MeSH Terms: conditions — Tuberculosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Group (Cases): 1. Subject aged 18 years of age or over
  2. Written, informed consent obtained.
  3. New diagnosis of tuberculosis and starting on anti-tuberculosis treatment
  4. Known diagnosis of diabetes or a raised IFCC HbA1c level (>= 48 mmol/mol) at the time of TB diagnosis
  Interventions: Diagnostic Test: TB Drug Levels
- Non-Diabetic Group (Controls): 1. Subject aged 18 years of age or over
  2. Written, informed consent obtained.
  3. New diagnosis of tuberculosis and starting on anti-tuberculosis treatment
  4. IFCC HbA1c level < 48mmol/mol and no known diagnosis of diabetes
  Interventions: Diagnostic Test: TB Drug Levels

INTERVENTIONS:
Diagnostic Test: TB Drug Levels — TB drug levels at 1-2 time points at weeks 2, 8 and 16

SUMMARY:
Diabetes significantly increases the risk of developing active tuberculosis (TB). Diabetic patients who do develop TB have worse treatment outcomes and overall mortality. TB also worsens blood glucose control in diabetics, the mechanism of which is not well understood. The incidence of type 2 diabetes is rising globally, and consequently diabetes and TB co-infection is increasingly common, and improving outcomes in this cohort is of growing importance.

Low TB drug levels in diabetic patients have been postulated as a reason for these worse outcomes. There is however contradictory evidence in the literature that TB drug levels really are consistently and significantly lower in diabetics compared with non-diabetics. If this were shown to be the case, performing therapeutic drug monitoring in diabetic patients may be a straightforward way to improve outcomes. Improving blood glucose control may also lead to improved outcomes, however there is nothing previously in the literature looking at detailed blood glucose monitoring in diabetic patients being treated for TB.

This study is planned as a case control study comparing 24 non-diabetic patients commencing TB treatment with 24 cases who have both TB and diabetes. Samples for post-dose TB drug levels will be taken at 2 time points at weeks 2, 8 and 16. These will be analysed via population pharmacokinetics to compare pharmacokinetic profiles between the 2 groups, with the hypothesis that the diabetic group will have a significantly lower exposure to TB drugs than the non-diabetic group. The diabetic group will also be asked to wear a continuous glucose monitor (blinded Dexcom) for 10 days at baseline and week 16, with data compared between the 2 time points.

DETAILED DESCRIPTION:
This study has been designed as a case control trial analysed via population pharmacokinetic modelling, with the hypothesis that overall exposure to TB medications will be lower in the diabetic than the non-diabetic group.

Non-Diabetic group (controls):

This group will be asked to take their TB medications as usual, and return at weeks 2 and 8 (timed to fit with routine appointments) and week 16. On these days, participants will be asked to record a video or to call the study team when taking the TB medications, so that the time can be recorded, and will then attend later in the day for routine bloods (week 2 and 8) and trial bloods taken at the same time (trial bloods only at week 16). At each visit, consent will be checked, the participant will be weighed and current medications will be checked. Venepuncture will be carried out for scheduled blood tests and for TB drug levels. With the participant's consent, a further blood sample will be taken later in the day for TB drug levels in addition.

Diabetic group (cases):

The diabetic group will undertake the same visits as the control group, with 2 additional features. Part of the same blood samples taken for TB drug levels will be used to measure oral diabetes drug levels in participants established on oral diabetes medication. These participants will be asked to attend an additional visit after the baseline visit but prior to starting TB treatment. Participants will be asked to record (again via video or call to the team) the time the evening diabetes medications were taken, to omit the morning dose and then to attend for a blood sample for a baseline diabetes medication level. Diabetic patient will also wear a blinded continuous glucose monitor (CGM) for 10 days at baseline and at week 16. Participants will be trained, and at weeks 0 and 16, the study co-ordinator will apply the sensor and transmitter, which will be worn for the next 10 days. The data will then be analysed to compare week 0 with week 16.

Corticosteroid Subgroup:

As a pilot project, any patients commencing on TB therapy who are also receiving corticosteroids as part of TB treatment, will be approached to follow the sample schedule as the control group.

Blood samples will be processed within 30 minutes of venepuncture, and the serum fraction (which contains the medications) will be frozen to -20C at the on-site laboratory. Frozen samples will be transported to the testing laboratory in appropriately labelled containers. Batches of samples will be analysed using high performance liquid chromatography for TB and diabetes drug levels.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Subject aged 18 years of age or over
* Written, informed consent obtained.
* New diagnosis of tuberculosis and starting on anti-tuberculosis treatment
* Known diagnosis of diabetes or a raised IFCC HbA1c level (>= 48 mmol/mol) at the time of TB diagnosis

Controls:

* Subject aged 18 years of age or over
* Written, informed consent obtained.
* New diagnosis of tuberculosis and starting on anti-tuberculosis treatment
* IFCC HbA1c level < 48mmol/mol and no known diagnosis of diabetes

Exclusion Criteria:

* Subject aged under 18 years
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from TB clinics at London North West University NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Rifampicin/Isoniazid/Pyrazinamide Cmax 2 hours post-dose | 2, 8, 16 weeks as discussed above
  To be measured via population pharmacokinetic modelling, with case group compared to control group.

SECONDARY OUTCOMES:
Antidiabetic medication Cmax at baseline and 2 hours post dose | Baseline, 2, 8 and 16 weeks as discussed above
  To be measured via population pharmacokinetic modelling, with baseline compared to weeks 2, 8 and 16.
Mean daily subcutaneous glucose measurement | Baseline and 16 weeks for 10 days each
  Via CGM comparing baseline with week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ann Sturdy, Principal Investigator — LONDON NORTH WEST UNIVERSITY HEALTHCARE NHS TRUST
Locations (1):
- London North West University NHS University Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided